CLINICAL TRIAL: NCT04137809
Title: TREAT Foot Drop After Stroke With Ankle Robot
Acronym: TREAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to logistical and safety concerns relating to Covid-19.
Sponsor: NextStep Robotics Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A-7010546431
Record Dates: First submitted 2019-10-11; First posted 2019-10-24 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Foot Drop; Stroke; Hemiparesis
MeSH Terms: conditions — Peroneal Neuropathies; Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot Group (Experimental): 1-arm study where eligible volunteers will undergo robotic testing for safety, comfort, and fit.
  Interventions: Device: AMBLE

INTERVENTIONS:
Device: AMBLE — Treadmill walking while wearing AMBLE device; three times a week for two weeks; 45-60 minutes per session.

SUMMARY:
Researchers at the University of Maryland Rehabilitation and Orthopaedic Institute are looking for individuals who have suffered a stroke and have leg and ankle weakness (foot-drop), to participate in a pilot study to examine the safety and effectiveness of an ankle robot walking program on walking function

This is the first in human test of walking training over-ground using a wearable, lightweight, battery operated ankle robot exoskeleton; with assistance by trained research personnel for safety. This exercise device is aimed at assisting the foot during walking to reduce foot drop and improve walking safety in chronic, mild to moderately impaired stroke survivors who have foot drop.

Possible risks of participating in this study are described in this document. The greatest risks include the risk of falling, muscle soreness, skin irritation, or cardiovascular complications. Before starting, you will have a medical history and medical assessments performed to determine if this study is safe for you. All sessions will be assisted by trained research personnel under supervision of a physical therapist, with medical personnel locally on call.

DETAILED DESCRIPTION:
This study is designed to see if the ankle robot is safe and effective to use in restoring gait function in individuals with foot drop.

This research project will be conducted at the University of Maryland Rehabilitation and Orthopaedic Institute (UM Rehab). There will be approximately 10 individuals from the Baltimore, Maryland area recruited to voluntarily participate in this study.

If you take part in this research, you will be asked:

* To participate in this study for approximately 10 weeks total.
* Attend at least 6 ankle robot gait training sessions that will last 45-60 minutes each session, 3 times a week for 2 weeks at UM Rehab.
* Undergo a medical and neurological evaluation at screening.
* Perform balance and walking tests with and without your usual assistive walking device.
* Walk on a treadmill with the ankle robot on your foot.
* Report to the research team any changes to assistive walking device usage between training sessions, and any health-related issues or changes.
* Maintain your current medications at their current doses and schedules throughout this study, or inform the study physician about any medication changes.
* Not to participate in any other study that would affect our results.
* You will be seated and fitted with the ankle robot before each testing visit and each gait training session. During the fitting process, the ankle robot will be secured to the stroke affected lower leg using a modified shin guard that has Velcro straps. Regular shoes will be worn. The "shoe covered" affected foot will be inserted into a modified slipper. Comfort and fit will be noted. Should you have any discomfort or feeling like the ankle robot device is rubbing on skin, padding will be applied to protect the skin.
* A gait belt will be worn around the waist and research staff will use this belt to provide support, and to protect against falls during the balance/walking tests and during ankle robot gait training sessions.
* Gait training sessions will be conducted with usual assistive devices for balance and with the ankle robot turned on and turned off.
* The research team will periodically collect heart rate and blood pressure measurements to determine how hard you are working during various tasks. You will be asked how you feel while performing these tasks. Researchers will use this information to guide the gait training program.

Tests will be completed at 3 points: baseline (before beginning training), after the 2-week gait training program, and then 6 weeks after the program.

* 3 tests of balance, mobility and gait.
* Timed walking tests (10 meter and 6-minute walks) to determine functional capacity with and without assistive walking devices, and with the ankle robot both turned on and turned off.
* Walking on a treadmill (wearing a safety harness) to assess walking patterns while wearing the ankle robot both turned on and turned off.
* Walking stability tests while wearing the ankle robot device both turned on and turned off. Usual assistive walking devices (cane or walker) will be used, if necessary. The testing tasks will be performed with and without your ankle foot orthosis, if one is worn.

In some instances, if sessions are canceled due to personal or other uncontrollable factors, time in the study may exceed 10 weeks. We do not expect time commitments to exceed 14 weeks.

If there are medical or other reasons that require time away from the study for more than one month, baseline tests will be repeated, and training will resume starting at session #1.

The investigator will ask if data can be collected from your routine medical care. If agreed upon, this data will be handled the same as research data.

If granted permission, we will photograph/videotape training sessions and test visits, to provide feedback on progress during the study.

There is an option to allow these photographs/recordings to be kept by the research team for use in future presentations (slideshows, conferences, etc.) and to educate others about this research study.

POTENTIAL RISKS/DISCOMFORTS:

This study exposes you to several risks:

* Skin irritation: There is a risk that wearing the ankle robot may cause skin irritation with repeated ankle movements. The research team will check skin before and after each training session for signs of skin redness or irritation. Foam padding will be used to provide protection to skin if needed. The padding will be adjusted if any discomfort develops during any training visits or testing sessions.
* Fall risk: Falls could occur during the gait training, balance or walking tests. We will reduce the likelihood of falling by having 2 research team members present at all sessions. One team member (spotter) will walk behind you providing support by holding onto the gait belt worn around the waist. The other team member will assist the spotter and will monitor the room for potential trip hazards. A safety harness will be worn to protect against falls during walking tests performed on the treadmill.
* Muscle discomfort: Muscle soreness may be experienced. This risk is greatest during the early stages of this study before familiarization with the study-related activities. We will monitor muscle soreness during and between sessions. We will address muscle soreness by adjusting training by providing more frequent or longer rest breaks. Muscle soreness will also be addressed by applying ice to sore muscles and teaching appropriate stretching exercises.
* Joint pain: There is a very slight risk that the robot could move the foot in the wrong direction, causing joint discomfort. This is extremely unlikely, as maximal force outputs by the robot are not sufficient to cause injury to a muscle, tendon, or ligament. Further protection is provided by fail-safe switches that quickly turn the robot off in 2 milliseconds. An engineer technician will perform service checks (calibration and operational) to the robot device before and after each session. We will address joint soreness by adjusting training by providing more frequent or longer rest breaks. Joint soreness will also be addressed by applying ice to sore regions.
* Cardiac risks: This ankle robot training program is considered low intensity exercise. Exercise training can be associated with the risk of cardiovascular complications such as chest pain, heart attack, or sudden death and complications related to stress and strains of muscles, twisted ankles, or falls. This risk is increased in people who have heart disease, poor circulation to the legs, or stroke. The risk of heart attack in these people is one in 300,000 hours of exercise, and risk of death is one in 800,000 hours of exercise.
* To minimize this risk, you will first undergo a medical evaluation. All walking training sessions will be supervised by personnel trained in cardiopulmonary resuscitation (CPR), and a clinical provider will be on call. Heart rate and blood pressure will be assessed by trained study team members before and after each training session or more frequently, if indicated.
* If blood pressure or heart rate go too high or an irregular heart rate, chest pain, or leg cramps develop, the training session will be stopped immediately. An AED (automatic external defibrillator) is available on site. A "rapid response" medical team will be contacted if a medical emergency occurs during a session. This team will evaluate a participant's condition and determine if they should be transported to the nearest hospital. Heart rate and blood pressure will be periodically monitored during each session. Instructions about warning signs of cardiac events will be given (for example: chest pain, shortness of breath, lightheadedness, and pain in the arms) and reminded about these symptoms during the study.
* Privacy and confidentiality: Research staff will collect personal information during this study. This information will be protected, however, we cannot be assured of absolute privacy. This data will be kept locked in the Rehabilitation Research Center at the University of Maryland Rehabilitation and Orthopaedic Institute (UM Rehab). Personal data (name, address, and other identifiers) will remain strictly confidential. Data will be coded to protect privacy. This coded data will be used in scientific publications and presentations, and will not be personally identified. The risk of loss confidentiality will be minimized by storing data, photos, and any recorded imaging in a secure location in a locked office within a locked cabinet, with access restricted to research staff.
* Unknown risks: In addition to the risks described in this form, there may be unknown mild risks/discomforts involved in participating in this study. The research staff will update you on any new information that may affect health, welfare, or decision to stay in the study.

POTENTIAL BENEFITS

There is no guarantee that a direct benefit from participation in this study will be received. Participation may help in the development of new robotic therapies for persons with foot drop, and to learn more about how to identify those who can successfully use this robotic approach to address their foot drop.

ALTERNATIVES TO PARTICIPATION

Participation is voluntary, and the alternative is not to participate. Conventional therapy may be an alternative to taking part in this study.

COSTS TO PARTICIPANTS

There will be no uncovered research-related costs. If you are injured because of study participation, you will receive emergency medical care if needed, and assistance in getting other medical care as needed. You or your carrier will be billed for the cost of care, just as you would be billed for any other medical care. It is not the University's policy to pay compensation to research subjects for injuries resulting from a study. The study staff can give more information about this if there is a study injury. Legal compensation for any injury that may occur during the study as a result of an error by a member of the research staff or by the sponsor may be sought.

RIGHT TO WITHDRAW

Participation in this study is voluntary. You are free to withdraw their consent at any time. Refusal to take part or to stop taking part in the study will involve no penalty or loss of benefits to which they are otherwise entitled. There are no other adverse consequences (physical, social, economic, legal, or psychological), if choosing to withdraw from the research.

REMOVAL FROM RESEARCH

The investigator or sponsor can decide to withdraw you from the study at any time without your approval. Removal from the study can be for reasons related solely to you, for example, not following study-related directions to related to research participation, a new treatment becomes available for foot drop, or a new medical illness occurs. Also, the research study may be stopped by the sponsor, the Investigator, or the Institutional Review Board. The research staff will discuss all details of a study withdrawal or the study closure with participants. Questions can be asked, should this happen. The sponsor may also decide to stop the Investigator's participation in the study. In that case, participation will end unless another investigator is identified and approved by the sponsor and the Institutional Review Board. Any significant new findings which develop during the study which may affect your willingness to participate in the study will be given.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75 years
* Greater than 3 months post stroke
* Hemiparetic stroke with foot drop (Dorsiflexion deficit)
* Dorsiflexion deficit for active range of motion (unable to reach zero degrees)
* Dorsiflexion deficit for strength with a manual motor score between 1/5 and 4/5
* Mild-moderate severity hemiparetic gait, identified by reduced stance, or reduced stance plus increased swing on affected side
* Able to participate in physical therapy for mobility recovery, defined by capacity to walk 10-m over-ground, albeit with minimal assist (FIM Mobility Subscale 4; subject can perform 75% of the task), supervision (FIM Mobility Score 5) or modified independence (FIM Mobility Score 6; use an assistive device)
* Adequate language and cognitive function to participate in routine mobility physical therapy

Exclusion Criteria:

* Cardiac history of unstable angina, recent (<3 mos.) myocardial infarction, congestive heart failure, significant valvular dysfunction
* Hypertension contraindicating rehabilitation (>160/100, two assessments)
* Peripheral arterial occlusive disease (Fontaine II)
* Orthopedic/chronic pain conditions precluding robot use
* Pulmonary or renal failure or active cancer
* Non-stroke neuromuscular or neurological conditions that restrict gait or could confound interpretation of key outcomes
* Aphasia, unable to follow 2 step commands, or communicate pain, discomfort, or sufficiently interact with PT/staff to participate in PT or PTR treatment assignments, as per judgment of a credentialed clinician
* Cognitive dysfunction that confounds participation, including diagnosis of dementia including Alzheimer's Disease and Alzheimer's Related Disorders, or active delirium (as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM- 5));
* Modified Ashworth Spasticity >3 (considerable increase in muscle tone, passive movement difficult) or contractures that preclude adequate volitional range of motion (ROM) for motor learning
* Foot and lower leg pain or deformities that complicate safe and effective robot fit
* Active deep venous thrombosis
* Skin lesions, infections, other cutaneous or musculoskeletal conditions of the shank that would complicate robot attachment to the leg
* Untreated and active major depression

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Participant report as to whether they are comfortable wearing the device while walking (5 point Likert Scale) | Change from Baseline at both 2 Weeks and at 8 Weeks
  The Likert questionnaire will consist of items related to self-reported measures of comfort including the presence of any abrasions on skin, musculoskeletal issues such as pain resulting from pinch points, and other issues related to overall discomfort.
10-meter Walk Test | Change from Baseline at both 2 Weeks and at 8 Weeks
  Time(seconds) is measured while the individual walks 10 meters.
6-minute Walk Test | Change from Baseline at both 2 Weeks and at 8 Weeks
  Assesses distance (meters) walked over 6 minutes.
Presence of Swing Plantar-flexion | Change from Baseline at both 2 Weeks and at 8 Weeks
  Number of subjects with swing plantar-flexion as assessed by a blinded physical therapist assessment through video recording.
Donning/Doffing Time | Baseline
  Average time (minutes) for donning/doffing the device per subject over the course of intervention.
Average Time of Use | Chang from Baseline at 2 Weeks
  Average time (hours) of device use per subject over the course of intervention.

SECONDARY OUTCOMES:
Berg Balance Scale | Change from Baseline at both 2 Weeks and at 8 Weeks
  A 14-item objective measure designed to assess static balance and fall risk; ranges from 0-56; higher score is better.
Dynamic Gait Index | Change from Baseline at both 2 Weeks and at 8 Weeks
  Assesses gait, balance, and fall risk; ranges from 0-24; higher score is better.
Swing Dorsiflexion | Change from Baseline at both 2 Weeks and at 8 Weeks
  Peak swing dorsiflexion averaged across each gait cycle for each subject at a given testing time point.
Angle at Initial Contact | Change from Baseline at both 2 Weeks and at 8 Weeks
  Angle at initial contact averaged across each gait cycle for each subject at a given testing time point.
Number of Heel-First Foot Strikes | Change from Baseline at both 2 Weeks and at 8 Weeks
  Number of heel-first foot strikes for each subject at a given testing time point.
Number of Participants Using Assistive Devices and Ankle Foot Orthoses | Change from Baseline at both 2 Weeks and at 8 Weeks
  Number of Participants Using Assistive Devices and Ankle Foot Orthoses.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Macko, MD, Principal Investigator — University of Maryland, College Park; Bradley Hennessie, MHA,MBA, Study Director — NextStep Robotics Inc.
Locations (1):
- UM Rehabilitation & Orthopaedic Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available immediately following any and all publications arising from the study.
Access Criteria: Publications can be accessed through journal websites and conference proceedings. This information will be made available to researchers and, more broadly, members of the public.

REFERENCES:
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Background] Forster A, Young J. Incidence and consequences of falls due to stroke: a systematic inquiry. BMJ. 1995 Jul 8;311(6997):83-6. doi: 10.1136/bmj.311.6997.83. PMID 7613406
- [Background] Ramnemark A, Nyberg L, Borssen B, Olsson T, Gustafson Y. Fractures after stroke. Osteoporos Int. 1998;8(1):92-5. doi: 10.1007/s001980050053. PMID 9692083
- [Background] Dennis MS, Lo KM, McDowall M, West T. Fractures after stroke: frequency, types, and associations. Stroke. 2002 Mar;33(3):728-34. doi: 10.1161/hs0302.103621. PMID 11872896
- [Background] Kanis J, Oden A, Johnell O. Acute and long-term increase in fracture risk after hospitalization for stroke. Stroke. 2001 Mar;32(3):702-6. doi: 10.1161/01.str.32.3.702. PMID 11239190
- [Background] Bosch PR, Harris JE, Wing K; American Congress of Rehabilitation Medicine (ACRM) Stroke Movement Interventions Subcommittee. Review of therapeutic electrical stimulation for dorsiflexion assist and orthotic substitution from the American Congress of Rehabilitation Medicine stroke movement interventions subcommittee. Arch Phys Med Rehabil. 2014 Feb;95(2):390-6. doi: 10.1016/j.apmr.2013.10.017. Epub 2013 Nov 6. PMID 24211493
- [Background] Bethoux F, Rogers HL, Nolan KJ, Abrams GM, Annaswamy T, Brandstater M, Browne B, Burnfield JM, Feng W, Freed MJ, Geis C, Greenberg J, Gudesblatt M, Ikramuddin F, Jayaraman A, Kautz SA, Lutsep HL, Madhavan S, Meilahn J, Pease WS, Rao N, Seetharama S, Sethi P, Turk MA, Wallis RA, Kufta C. Long-Term Follow-up to a Randomized Controlled Trial Comparing Peroneal Nerve Functional Electrical Stimulation to an Ankle Foot Orthosis for Patients With Chronic Stroke. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):911-22. doi: 10.1177/1545968315570325. Epub 2015 Feb 4. PMID 25653225
- [Background] Sheffler LR, Bailey SN, Wilson RD, Chae J. Spatiotemporal, kinematic, and kinetic effects of a peroneal nerve stimulator versus an ankle foot orthosis in hemiparetic gait. Neurorehabil Neural Repair. 2013 Jun;27(5):403-10. doi: 10.1177/1545968312465897. Epub 2012 Nov 27. PMID 23192416
- [Background] Ring H, Treger I, Gruendlinger L, Hausdorff JM. Neuroprosthesis for footdrop compared with an ankle-foot orthosis: effects on postural control during walking. J Stroke Cerebrovasc Dis. 2009 Jan;18(1):41-7. doi: 10.1016/j.jstrokecerebrovasdis.2008.08.006. PMID 19110144
- [Background] Kluding PM, Dunning K, O'Dell MW, Wu SS, Ginosian J, Feld J, McBride K. Foot drop stimulation versus ankle foot orthosis after stroke: 30-week outcomes. Stroke. 2013 Jun;44(6):1660-9. doi: 10.1161/STROKEAHA.111.000334. Epub 2013 May 2. PMID 23640829
- [Background] Everaert DG, Stein RB, Abrams GM, Dromerick AW, Francisco GE, Hafner BJ, Huskey TN, Munin MC, Nolan KJ, Kufta CV. Effect of a foot-drop stimulator and ankle-foot orthosis on walking performance after stroke: a multicenter randomized controlled trial. Neurorehabil Neural Repair. 2013 Sep;27(7):579-91. doi: 10.1177/1545968313481278. Epub 2013 Apr 4. PMID 23558080
- [Background] Nair PM, Rooney KL, Kautz SA, Behrman AL. Stepping with an ankle foot orthosis re-examined: a mechanical perspective for clinical decision making. Clin Biomech (Bristol). 2010 Jul;25(6):618-22. doi: 10.1016/j.clinbiomech.2010.03.001. Epub 2010 Apr 1. PMID 20362373
- [Background] Burdett RG, Borello-France D, Blatchly C, Potter C. Gait comparison of subjects with hemiplegia walking unbraced, with ankle-foot orthosis, and with Air-Stirrup brace. Phys Ther. 1988 Aug;68(8):1197-203. PMID 3399515
- [Background] Radtka SA, Oliveira GB, Lindstrom KE, Borders MD. The kinematic and kinetic effects of solid, hinged, and no ankle-foot orthoses on stair locomotion in healthy adults. Gait Posture. 2006 Oct;24(2):211-8. doi: 10.1016/j.gaitpost.2005.09.005. Epub 2005 Nov 2. PMID 16260141
- [Background] Forrester LW, Roy A, Hafer-Macko C, Krebs HI, Macko RF. Task-specific ankle robotics gait training after stroke: a randomized pilot study. J Neuroeng Rehabil. 2016 Jun 2;13(1):51. doi: 10.1186/s12984-016-0158-1. PMID 27255156
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Feigin VL, Roth GA, Naghavi M, Parmar P, Krishnamurthi R, Chugh S, Mensah GA, Norrving B, Shiue I, Ng M, Estep K, Cercy K, Murray CJL, Forouzanfar MH; Global Burden of Diseases, Injuries and Risk Factors Study 2013 and Stroke Experts Writing Group. Global burden of stroke and risk factors in 188 countries, during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet Neurol. 2016 Aug;15(9):913-924. doi: 10.1016/S1474-4422(16)30073-4. Epub 2016 Jun 9. PMID 27291521
- [Background] Neptune RR, Kautz SA, Zajac FE. Contributions of the individual ankle plantar flexors to support, forward progression and swing initiation during walking. J Biomech. 2001 Nov;34(11):1387-98. doi: 10.1016/s0021-9290(01)00105-1. PMID 11672713
- [Background] Bowden MG, Balasubramanian CK, Neptune RR, Kautz SA. Anterior-posterior ground reaction forces as a measure of paretic leg contribution in hemiparetic walking. Stroke. 2006 Mar;37(3):872-6. doi: 10.1161/01.STR.0000204063.75779.8d. Epub 2006 Feb 2. PMID 16456121
- [Background] Olney SJ, Griffin MP, Monga TN, McBride ID. Work and power in gait of stroke patients. Arch Phys Med Rehabil. 1991 Apr;72(5):309-14. PMID 2009047
- [Background] Gersten JW, Orr W. External work of walking in hemiparetic patients. Scand J Rehabil Med. 1971;3(1):85-8. No abstract available. PMID 5156160
- [Background] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Management of Stroke Rehabilitation Working Group. VA/DOD Clinical practice guideline for the management of stroke rehabilitation. J Rehabil Res Dev. 2010;47(9):1-43. No abstract available. PMID 21213454
- [Background] Wagner TH, Lo AC, Peduzzi P, Bravata DM, Huang GD, Krebs HI, Ringer RJ, Federman DG, Richards LG, Haselkorn JK, Wittenberg GF, Volpe BT, Bever CT, Duncan PW, Siroka A, Guarino PD. An economic analysis of robot-assisted therapy for long-term upper-limb impairment after stroke. Stroke. 2011 Sep;42(9):2630-2. doi: 10.1161/STROKEAHA.110.606442. Epub 2011 Jul 14. PMID 21757677
- [Background] Hogan N. Impedance Control: An Approach to Manipulation: Part I-Theory. ASME. J. Dyn. Sys., Meas., Control. 1985;107(1):1-7.
- [Background] Olney SJ, Richards C. Hemiparetic gait following stroke. Part I: Characteristics. Gait Posture. 1996; 4:136-48.
- [Background] Roy A, Krebs HI, Williams DJ, Bever CT, Forrester LW, Macko RF, Hogan N. Robot-aided neurorehabilitation: a robot for ankle rehabilitation. IEEE Trans Robotics. 2009; 25:569-82
- [Background] Hogan N. Impedance Control: An Approach to Manipulation: Part II-Implementation. ASME. J. Dyn. Sys., Meas., Control. 1985;107(1):8-16
- [Background] Hogan N. Impedance Control: An Approach to Manipulation: Part III-Applications. ASME. J. Dyn. Sys., Meas., Control. 1985;107(1):17-24.
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Kendall FP, McCreary EK, Provance PG, Rodgers MM, Romani WA. Muscles: Testing and function with posture and pain, 5th edition, 2005, Lippincott Williams & Wilkins, Baltimore, MD
- [Background] Norkin C, White D. Measurement of joint motion: A guide to goniometry, 3rd edition, 2003, FA Davis, Philadelphia, PA.
- [Background] Butland RJ, Pang J, Gross ER, Woodcock AA, Geddes DM. Two-, six-, and 12-minute walking tests in respiratory disease. Br Med J (Clin Res Ed). 1982 May 29;284(6329):1607-8. doi: 10.1136/bmj.284.6329.1607. No abstract available. PMID 6805625
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547
- [Background] Jonsdottir J, Cattaneo D. Reliability and validity of the dynamic gait index in persons with chronic stroke. Arch Phys Med Rehabil. 2007 Nov;88(11):1410-5. doi: 10.1016/j.apmr.2007.08.109. PMID 17964880
- [Background] Forrester LW, Roy A, Goodman RN, Rietschel J, Barton JE, Krebs HI, Macko RF. Clinical application of a modular ankle robot for stroke rehabilitation. NeuroRehabilitation. 2013;33(1):85-97. doi: 10.3233/NRE-130931. PMID 23949045
- [Background] Forrester LW, Roy A, Krywonis A, Kehs G, Krebs HI, Macko RF. Modular ankle robotics training in early subacute stroke: a randomized controlled pilot study. Neurorehabil Neural Repair. 2014 Sep;28(7):678-87. doi: 10.1177/1545968314521004. Epub 2014 Feb 10. PMID 24515923
- [Background] Forrester LW, Roy A, Krebs HI, Macko RF. Ankle training with a robotic device improves hemiparetic gait after a stroke. Neurorehabil Neural Repair. 2011 May;25(4):369-77. doi: 10.1177/1545968310388291. Epub 2010 Nov 29. PMID 21115945
- [Background] Roy A, Krebs HI, Bever CT, Forrester LW, Macko RF, Hogan N. Measurement of passive ankle stiffness in subjects with chronic hemiparesis using a novel ankle robot. J Neurophysiol. 2011 May;105(5):2132-49. doi: 10.1152/jn.01014.2010. Epub 2011 Feb 23. PMID 21346215
- [Background] Ovbiagele B, Goldstein LB, Higashida RT, Howard VJ, Johnston SC, Khavjou OA, Lackland DT, Lichtman JH, Mohl S, Sacco RL, Saver JL, Trogdon JG; American Heart Association Advocacy Coordinating Committee and Stroke Council. Forecasting the future of stroke in the United States: a policy statement from the American Heart Association and American Stroke Association. Stroke. 2013 Aug;44(8):2361-75. doi: 10.1161/STR.0b013e31829734f2. Epub 2013 May 22. PMID 23697546
- [Background] Macko RF, Ivey FM, Forrester LW, Hanley D, Sorkin JD, Katzel LI, Silver KH, Goldberg AP. Treadmill exercise rehabilitation improves ambulatory function and cardiovascular fitness in patients with chronic stroke: a randomized, controlled trial. Stroke. 2005 Oct;36(10):2206-11. doi: 10.1161/01.STR.0000181076.91805.89. Epub 2005 Sep 8. PMID 16151035
- [Background] Macko RF, DeSouza CA, Tretter LD, Silver KH, Smith GV, Anderson PA, Tomoyasu N, Gorman P, Dengel DR. Treadmill aerobic exercise training reduces the energy expenditure and cardiovascular demands of hemiparetic gait in chronic stroke patients. A preliminary report. Stroke. 1997 Feb;28(2):326-30. doi: 10.1161/01.str.28.2.326. PMID 9040684
- [Background] Macko RF, Ivey FM, Forrester LW. Task-oriented aerobic exercise in chronic hemiparetic stroke: training protocols and treatment effects. Top Stroke Rehabil. 2005 Winter;12(1):45-57. doi: 10.1310/PJQN-KAN9-TTVY-HYQH. PMID 15736000
- [Background] Goodman RN, Rietschel JC, Roy A, Jung BC, Diaz J, Macko RF, Forrester LW. Increased reward in ankle robotics training enhances motor control and cortical efficiency in stroke. J Rehabil Res Dev. 2014;51(2):213-27. doi: 10.1682/JRRD.2013.02.0050. PMID 24933720
- [Background] Roy A, Forrester LW, Macko RF. Short-term ankle motor performance with ankle robotics training in chronic hemiparetic stroke. J Rehabil Res Dev. 2011;48(4):417-29. doi: 10.1682/jrrd.2010.04.0078. PMID 21674391
- [Background] Roy A, Krebs HI, Barton JE, Macko RF, Forrester LW. Anklebot-assisted locomotor training after stroke: A novel deficit-adjusted control approach. In: Proc 2013 IEEE Int. Conf Rob Auto (ICRA). 2013; 2175-82.
- [Background] Roy A, Forrester LW, Macko F. Method and apparatus for providing deficit-adjusted adaptive assistance during movement phases of an impaired joint. US Patent 9,943,459, filed November 20, 2014, and issued April 17, 2018.
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] National Institute of Health, National Institute of Neurological Disorders and Stroke. Stroke Scale. http://www.ninds.nih.gov/doctors/NIH_Stroke_Scale.pdf
- [Background] Devins, G. M., & Orme, C. M. Center for epidemiologic studies depression scale. Test critiques. 1985; 2: 144-60.
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Background] Shumway-Cook A, Woollacott MH. Motor control: Theory and practical applications, 2nd Edition, 2001, Baltimore: Lippincott Williams and Wilkins
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Tinetti ME, Mendes de Leon CF, Doucette JT, Baker DI. Fear of falling and fall-related efficacy in relationship to functioning among community-living elders. J Gerontol. 1994 May;49(3):M140-7. doi: 10.1093/geronj/49.3.m140. PMID 8169336
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Buck D, Jacoby A, Massey A, Steen N, Sharma A, Ford GA. Development and validation of NEWSQOL, the Newcastle Stroke-Specific Quality of Life Measure. Cerebrovasc Dis. 2004;17(2-3):143-52. doi: 10.1159/000075783. Epub 2003 Dec 23. PMID 14707414
- [Background] Little RJA, Rubin DB. Statistical analysis with missing data. 1987
- [Background] Armitage P, Berry G, Matthews JNS. Statistical methods in medical research. 2002;4th edition